CLINICAL TRIAL: NCT03915496
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP, MULTI-CENTER STUDY TO INVESTIGATE THE MECHANISM OF ACTION OF ABROCITINIB MONOTHERAPY IN ADULT PARTICIPANTS WITH MODERATE-TO-SEVERE ATOPIC DERMATITIS
Brief Title: Study Evaluating the Mechanism of Action of PF-04965842 Monotherapy for Moderate-to-severe Atopic Dermatitis
Acronym: JADE MOA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451037; JADE MOA (Other: Alias Study Number)
Record Dates: First submitted 2019-03-22; First posted 2019-04-16 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; atopic eczema; eczema; JAK; janus kinase
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-04965842 200 mg (Experimental)
  Interventions: Drug: PF-04965842 200 mg
- PF-04965842 100 mg (Experimental)
  Interventions: Drug: PF-04965842 100 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04965842 200 mg — PF-04965842 200 mg administered as two tablets to be taken orally once daily for 12 weeks
  Arms: PF-04965842 200 mg
Drug: PF-04965842 100 mg — PF-04965842 100 mg administered as two tablets to be taken orally once daily for 12 weeks
  Arms: PF-04965842 100 mg
Drug: Placebo — Placebo administered as two tablets to be taken orally once daily for 12 weeks
  Arms: Placebo

SUMMARY:
B7451037 is a randomized, double-blind, placebo-controlled, parallel-group, Phase 2a study to investigate the mechanism of action of PF-04965842 by correlating efficacy outcomes with changes from baseline in key skin and blood biomarkers in adult participants at least 18 years of age with moderate-to-severe atopic dermatitis. Participants will be screened within 28 days prior to the first dose of study intervention to confirm eligibility. A total of approximately 51 participants will be randomized in a 1:1:1 ratio to receive PF-04965842 200 mg once daily (QD), PF004965842 100 mg QD, or matching placebo QD for 12 weeks. At the end of the 12-week study treatment, qualified participants will have the option to enter the long-term extension study B7451015 (NCT03422822). Participants discontinuing early from this study will undergo a 4-week off-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic moderate-to-severe atopic dermatitis (AD) for at least 1 year
* Recent history of inadequate response to medicated topical therapy for AD or required systemic therapy to control disease
* Moderate-to-severe AD defined as affected BSA at least 10%, IGA at least 3, EASI at least 16, Peak Pruritus NRS at least 4

Exclusion Criteria:

* A current or past medical history of conditions associated with thrombocytopenia, coagulopathy, or platelet dysfunction
* Currently have active forms of other inflammatory skin diseases, i.e. not AD, or have evidence of skin conditions (e.g. psoriasis, seborrheic dermatitis, lupus) at the time of Day 1 that would interfere with evaluation of AD or response to treatment
* Participants who have received prior treatment with any systemic JAK inhibitors
* Require treatment with prohibited concomitant medication(s) or have received a prohibited concomitant medication within specified time frames prior to the first dose of study medication, including topical treatments that could affect AD
* Pregnant or breastfeeding women or sexually-active women of childbearing potential who are unwilling to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (9):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Keck School of Medicine of USC - IDS Pharmacy, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Olympian Clinical Research, Largo, Florida
  - ForCare Clinical Research, Tampa, Florida
  - The Indiana Clinical Trials Center, PC - Dermatology Research, Plainfield, Indiana
  - Wayne Health - Wayne State Dermatology, Dearborn, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Menter Dermatology Research Institute, Dallas, Texas
- Canada (2):
  - Beacon Dermatology, Calgary, Alberta
  - Innovaderm Research, Inc., Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 adult participants with moderate-to-severe atopic dermatitis (AD) were randomized to the study and received study intervention, including 16 participants in the abrocitinib (PF-04965842) 100 mg once daily (QD) group, 14 participants in the abrocitinib 200 mg QD group, and 16 participants in the placebo group.
Groups:
- Abrocitinib 100 mg QD: Adult participants with moderate-to-severe AD received abrocitinib 100 mg QD for 12 weeks.
- Abrocitinib 200 mg QD: Adult participants with moderate-to-severe AD received abrocitinib 200 mg QD for 12 weeks.
- Placebo: Adult participants with moderate-to-severe AD received placebo QD for 12 weeks.
Period: Overall Study
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Started | 16 | 14 | 16
Completed | 14 | 13 | 14
Not Completed | 2 | 1 | 2
Not completed — Adverse Event | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (19.41) | 41.4 (16.72) | 38.9 (15.64) | 42.4 (17.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 3 | 21
  Male | 5 | 7 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 8
  Not Hispanic or Latino | 13 | 12 | 11 | 36
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 10 | 5 | 11 | 26
  Black or African American | 4 | 1 | 2 | 7
  Asian | 1 | 6 | 2 | 9
  Multiracial | 0 | 1 | 1 | 2
  Not reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Fold-Change From Baseline in Atopic Dermatitis Biomarkers in Lesional and Non-lesional Skin at Week 12
Description: Mean fold-changes from baseline at Week 12 in the biomarkers for general inflammation (Matrix Metallopeptidase [MMP]12), hyperplasia (Keratin [KRT]16), Th2 immune response (C-C motif chemokine ligand [CCL]17, CCL18, CCL26), and Th22 immune response (S100 calcium binding protein A [S100A]8, S100A9, S100A12), in lesional (LS) and non-lesional (NL) skin tissues, respectively. Expression levels from RT-PCR are normalized to the housekeeping gene RPLP0 by negatively transforming the Ct values to -dCt.
Time Frame: Baseline, Week 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number Analyzed in each row refers to the number of participants measured and analyzed for each parameter at Week 12 visit.
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Fold change
  CCL17 (LS): number analyzed (Participants) | 14 | 13 | 13
  CCL17 (LS) | -5.896 (16.0867) | -15.604 (38.5469) | -0.729 (4.0821)
  CCL17 (NL): number analyzed (Participants) | 2 | 2 | 5
  CCL17 (NL) | -0.506 (7.5268) | -3.150 (2.6554) | -3.354 (7.6800)
  CCL18 (LS): number analyzed (Participants) | 14 | 13 | 13
  CCL18 (LS) | -11.600 (18.9748) | -24.558 (46.2466) | -1.096 (3.6800)
  CCL18 (NL): number analyzed (Participants) | 2 | 2 | 5
  CCL18 (NL) | -18.307 (24.0808) | -12.328 (13.3680) | -0.761 (2.8516)
  CCL26 (LS): number analyzed (Participants) | 14 | 13 | 13
  CCL26 (LS) | -3.886 (9.6426) | -0.464 (5.2150) | -0.205 (1.7928)
  CCL26 (NL): number analyzed (Participants) | 2 | 2 | 5
  CCL26 (NL) | -3.619 (2.1674) | -4.369 (8.0621) | 0.026 (2.0613)
  KRT16 (LS): number analyzed (Participants) | 14 | 13 | 13
  KRT16 (LS) | -24.604 (47.3896) | -53.285 (70.6935) | -1.898 (19.4730)
  KRT16 (NL): number analyzed (Participants) | 2 | 2 | 5
  KRT16 (NL) | -3.179 (6.2518) | -2.947 (1.4188) | -2.674 (7.2836)
  MMP-12 (LS): number analyzed (Participants) | 14 | 13 | 13
  MMP-12 (LS) | -44.200 (123.0708) | -306.161 (503.8312) | -0.184 (3.0962)
  MMP-12 (NL): number analyzed (Participants) | 2 | 2 | 5
  MMP-12 (NL) | -20.822 (31.5640) | -27.523 (16.5608) | -1.897 (3.6968)
  S100A12 (LS): number analyzed (Participants) | 14 | 13 | 13
  S100A12 (LS) | -13.931 (23.9740) | -1322.88 (4594.187) | 5.994 (57.0002)
  S100A12 (NL): number analyzed (Participants) | 2 | 2 | 5
  S100A12 (NL) | 4.052 (0.4124) | -4.300 (4.2217) | -14.200 (21.2222)
  S100A8 (LS): number analyzed (Participants) | 14 | 13 | 13
  S100A8 (LS) | -76.158 (181.1015) | -312.430 (395.0796) | 1.213 (31.0236)
  S100A8 (NL): number analyzed (Participants) | 2 | 2 | 5
  S100A8 (NL) | -3.797 (3.9226) | -14.249 (13.2540) | -8.394 (10.7181)
  S100A9 (LS): number analyzed (Participants) | 14 | 13 | 13
  S100A9 (LS) | -52.132 (113.0256) | -304.023 (376.0106) | -2.136 (17.2326)
  S100A9 (NL): number analyzed (Participants) | 2 | 2 | 5
  S100A9 (NL) | -2.781 (5.6012) | -34.776 (42.4019) | -7.368 (10.0856)

2. Secondary Outcome: Fold-Change From Baseline in Cellular (T-cell and Dendritic Cell) Inflammation Markers at Week 12
Description: Mean fold-changes from baseline in immunohistochemistry analysis in lesional skin endpoints at Week 12 are presented. Fold-changes are computed by obtaining the antilog of log2 fold-changes, retaining the sign for log2 fold-change.
Time Frame: Baseline, Week 12
Population: The analysis population included all participants randomly assigned to study interventionand who took at least 1 dose of study intervention. Number Analyzed refers to the numberof participants evaluable for each category.
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Fold change
  CD11C | -1.622 [-2.404 to -1.094] | -2.460 [-3.719 to -1.627] | -1.326 [-1.968 to 1.118]
  CD3 | -1.952 [-2.979 to -1.279] | -2.371 [-3.696 to -1.521] | -1.054 [-1.610 to 1.450]
  Fc Epsilon R1 | -1.610 [-2.276 to -1.140] | -2.088 [-3.003 to -1.453] | 1.092 [-1.295 to 1.545]
  Macrophage mannose receptor 1 | -1.249 [-1.538 to -1.015] | -1.835 [-2.282 to -1.476] | -1.155 [-1.422 to 1.066]

3. Secondary Outcome: Fold-Change From Baseline in Epidermal Hyperplasia Markers in Skin Biopsies and Skin Thickness at Week 12
Description: Mean fold-changes from baseline in hyperplasia markers in skin biopsies at Week 12 are presented. Fold-changes are computed by obtaining the antilog of log2 fold-changes, retaining the sign for log2 fold-change.
Time Frame: Baseline, Week 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number Analyzed refers to the number of participants evaluable for each category.
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Fold change
  Ki-67 | -1.638 [-2.859 to 1.066] | -1.911 [-3.432 to -1.064] | -1.153 [-2.016 to 1.516]
  Thickness | -1.310 [-1.735 to 1.010] | -1.508 [-2.024 to -1.123] | -1.185 [-1.570 to 1.118]

4. Secondary Outcome: Fold-Change From Baseline in Blood Biomarkers for Inflammation and Immune Response at Week 12
Description: OLINK Proteomics Microassay was used to analyze biomarkers in serum to assess the effect of abrocitinib on the blood biomarkers. Mean fold-changes at Week 12 from baseline are listed. Baseline is defined as the last observation on or prior to day of first dose (Day 1).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Fold change
  C-C motif chemokine ligand 23 (CCL23): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 23 (CCL23) | -0.247 (0.3367) | -0.519 (0.3958) | -0.245 (0.4302)
  C-C motif chemokine ligand 17 (CCL17): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 17 (CCL17) | -0.619 (0.8281) | -0.880 (1.0630) | 0.108 (0.8299)
  Selectin E (SELE): number analyzed (Participants) | 14 | 14 | 14
  Selectin E (SELE) | -0.520 (0.6198) | -0.717 (0.6172) | -0.170 (0.3571)
  Integrin subunit beta 2 (ITGB2): number analyzed (Participants) | 14 | 14 | 14
  Integrin subunit beta 2 (ITGB2) | -0.280 (0.3067) | -0.574 (0.2649) | 0.058 (0.1877)
  Platelet-derived growth factor (PDGF) subunit B: number analyzed (Participants) | 14 | 14 | 14
  Platelet-derived growth factor (PDGF) subunit B | -0.057 (0.2185) | -0.182 (0.3561) | 0.085 (0.2916)
  PDGF subunit A: number analyzed (Participants) | 14 | 14 | 14
  PDGF subunit A | -0.360 (0.3354) | -0.590 (0.3884) | -0.039 (0.1802)
  Linker for activation of T cells (LAT): number analyzed (Participants) | 14 | 14 | 14
  Linker for activation of T cells (LAT) | -0.127 (0.4281) | -0.322 (0.3329) | -0.169 (0.3493)
  C-C motif chemokine ligand 24 (CCL24): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 24 (CCL24) | -0.283 (0.5321) | -0.342 (0.2439) | -0.191 (0.2425)
  Lipoprotein lipase (LPL): number analyzed (Participants) | 14 | 14 | 14
  Lipoprotein lipase (LPL) | -0.037 (0.5906) | 0.281 (0.7465) | -0.224 (0.7340)
  Interferon (IFN)-gamma: number analyzed (Participants) | 14 | 14 | 14
  Interferon (IFN)-gamma | 0.264 (1.2382) | 0.903 (1.9580) | 0.763 (1.1019)
  Interleukin 2 receptor subunit alpha (IL2-RA): number analyzed (Participants) | 14 | 14 | 14
  Interleukin 2 receptor subunit alpha (IL2-RA) | -0.852 (0.6237) | -0.921 (0.4530) | -0.219 (0.3161)
  Interleukin (IL)-1 alpha: number analyzed (Participants) | 14 | 14 | 14
  Interleukin (IL)-1 alpha | 0.118 (0.4804) | -0.114 (0.2527) | 0.046 (0.3275)
  C-C motif chemokine ligand 25 (CCL25): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 25 (CCL25) | 0.229 (0.3299) | 0.324 (0.4351) | 0.149 (0.2235)
  C-C motif chemokine ligand 28 (CCL28): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 28 (CCL28) | 0.014 (0.2452) | 0.108 (0.2932) | 0.011 (0.2962)
  C-C motif chemokine ligand 20 (CCL20): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 20 (CCL20) | -0.465 (1.1905) | 0.111 (0.8023) | -0.333 (0.6612)
  C-C motif chemokine ligand 19 (CCL19): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 19 (CCL19) | -0.653 (0.6620) | -1.217 (0.9084) | -0.012 (0.5347)
  C-C motif chemokine ligand 16 (CCL16): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 16 (CCL16) | -0.258 (0.2716) | -0.313 (0.1866) | -0.103 (0.2040)
  C-C motif chemokine ligand 11 (CCL11): number analyzed (Participants) | 14 | 14 | 14
  C-C motif chemokine ligand 11 (CCL11) | 0.030 (0.2617) | 0.109 (0.2891) | 0.060 (0.2005)
  MMP-12: number analyzed (Participants) | 14 | 14 | 14
  MMP-12 | -0.554 (0.9534) | -0.756 (0.6576) | -0.631 (0.9298)
  Tumor necrosis factor receptor superfamily member 9 (TNFRSF9): number analyzed (Participants) | 14 | 14 | 14
  Tumor necrosis factor receptor superfamily member 9 (TNFRSF9) | -0.437 (0.3796) | -0.608 (0.2665) | -0.136 (0.2562)
  Tumor necrosis factor receptor superfamily member 12A (TNFRSF12A): number analyzed (Participants) | 14 | 14 | 14
  Tumor necrosis factor receptor superfamily member 12A (TNFRSF12A) | -0.143 (0.3348) | -0.048 (0.3744) | -0.078 (0.4294)
  Matrix metalloproteinase-1 (MMP-1): number analyzed (Participants) | 14 | 14 | 14
  Matrix metalloproteinase-1 (MMP-1) | -0.118 (0.1546) | 0.004 (0.2445) | -0.002 (0.1309)
  Interleukin 20 receptor subunit alpha (IL-20RA): number analyzed (Participants) | 14 | 14 | 14
  Interleukin 20 receptor subunit alpha (IL-20RA) | 0.089 (0.2394) | -0.111 (0.2573) | -0.040 (0.2018)
  IL-18: number analyzed (Participants) | 14 | 14 | 14
  IL-18 | -0.488 (0.4737) | -0.578 (0.3460) | -0.182 (0.4037)
  IL-16: number analyzed (Participants) | 14 | 14 | 14
  IL-16 | -0.512 (0.5606) | -0.697 (0.5642) | -0.222 (0.5656)
  IL-12: number analyzed (Participants) | 14 | 14 | 14
  IL-12 | -0.548 (0.5020) | -0.628 (0.3935) | -0.141 (0.3341)
  IL-12B: number analyzed (Participants) | 14 | 14 | 14
  IL-12B | -0.560 (0.4540) | -0.637 (0.3808) | -0.059 (0.3230)
  IL-17C: number analyzed (Participants) | 14 | 14 | 14
  IL-17C | -0.250 (1.2265) | 0.136 (0.5533) | -0.784 (1.0808)
  IL-7: number analyzed (Participants) | 14 | 14 | 14
  IL-7 | -0.082 (0.4541) | -0.425 (0.5173) | -0.020 (0.5239)
  IL-27: number analyzed (Participants) | 14 | 14 | 14
  IL-27 | -0.099 (0.1617) | -0.177 (0.2611) | -0.073 (0.2250)
  IL-13: number analyzed (Participants) | 14 | 14 | 14
  IL-13 | -0.230 (0.4810) | -0.490 (0.6399) | -0.213 (0.6765)
  IL-17D: number analyzed (Participants) | 14 | 14 | 14
  IL-17D | 0.057 (0.3222) | -0.222 (0.2921) | -0.105 (0.2420)
  IL-20: number analyzed (Participants) | 14 | 14 | 14
  IL-20 | -0.155 (0.2843) | -0.171 (0.2315) | -0.137 (0.3877)
  IL-4: number analyzed (Participants) | 14 | 14 | 14
  IL-4 | -0.130 (0.6704) | -0.308 (0.5324) | -0.128 (0.3287)
  IL-4RA: number analyzed (Participants) | 14 | 14 | 14
  IL-4RA | -0.075 (0.2436) | -0.619 (0.7577) | -0.340 (0.5764)
  IL-2: number analyzed (Participants) | 14 | 14 | 14
  IL-2 | 0.005 (0.1927) | -0.069 (0.2345) | 0.050 (0.3024)
  IL-8: number analyzed (Participants) | 14 | 14 | 14
  IL-8 | 0.080 (0.8463) | 0.090 (0.8062) | 0.152 (0.9180)
  IL-5: number analyzed (Participants) | 14 | 14 | 14
  IL-5 | 0.049 (0.2578) | -0.164 (0.3214) | -0.020 (0.3306)
  IL-6: number analyzed (Participants) | 14 | 14 | 14
  IL-6 | -0.086 (0.9560) | 0.150 (1.4005) | -0.228 (1.1986)
  IL-10: number analyzed (Participants) | 14 | 14 | 14
  IL-10 | -0.180 (0.4616) | -0.087 (0.4255) | -0.182 (0.6735)
  IL-33: number analyzed (Participants) | 14 | 14 | 14
  IL-33 | 0.022 (0.2275) | -0.116 (0.2353) | -0.138 (0.2815)
  Cluster of differentiation (CD) 5: number analyzed (Participants) | 14 | 14 | 14
  Cluster of differentiation (CD) 5 | -0.373 (0.2546) | -0.405 (0.1488) | -0.064 (0.1640)
  CD4: number analyzed (Participants) | 14 | 14 | 14
  CD4 | -0.252 (0.3139) | -0.406 (0.2184) | -0.159 (0.3220)
  CD40: number analyzed (Participants) | 14 | 14 | 14
  CD40 | -0.049 (0.1755) | -0.065 (0.3002) | 0.039 (0.2065)
  Peptidase Inhibitor 3 (PI3): number analyzed (Participants) | 14 | 14 | 14
  Peptidase Inhibitor 3 (PI3) | -0.463 (0.6634) | -0.332 (0.6725) | -0.583 (0.8686)
  Tumor necrosis factor (TNF): number analyzed (Participants) | 14 | 14 | 14
  Tumor necrosis factor (TNF) | -0.328 (0.3560) | -0.227 (0.6622) | 0.036 (0.9515)
  C-X-C motif chemokine ligand 5 (CXCL5): number analyzed (Participants) | 14 | 14 | 14
  C-X-C motif chemokine ligand 5 (CXCL5) | -0.208 (0.2889) | -0.364 (0.4082) | 0.068 (0.4028)
  X-C motif chemokine ligand 1 (XCL1): number analyzed (Participants) | 14 | 14 | 14
  X-C motif chemokine ligand 1 (XCL1) | -0.540 (0.4209) | -0.897 (0.4253) | -0.051 (0.3028)
  Thymic stromal lymphopoietin (TSLP): number analyzed (Participants) | 14 | 14 | 14
  Thymic stromal lymphopoietin (TSLP) | -0.100 (0.4871) | -0.047 (0.5610) | 0.019 (0.4495)
  CXCL10: number analyzed (Participants) | 14 | 14 | 14
  CXCL10 | -0.268 (0.9825) | -0.549 (0.9508) | 0.363 (0.4782)
  CXCL11: number analyzed (Participants) | 14 | 14 | 14
  CXCL11 | -0.399 (0.6089) | -0.695 (0.7402) | 0.210 (0.4335)
  CXCL9: number analyzed (Participants) | 14 | 14 | 14
  CXCL9 | -0.161 (0.6273) | -0.406 (0.9061) | 0.159 (0.5395)
  CXCL1: number analyzed (Participants) | 14 | 14 | 14
  CXCL1 | -0.218 (0.3795) | -0.375 (0.3356) | -0.062 (0.3892)
  CXCL16: number analyzed (Participants) | 14 | 14 | 14
  CXCL16 | 0.031 (0.2575) | -0.033 (0.2503) | -0.011 (0.1563)
  Transforming growth factor (TGF)-beta-1: number analyzed (Participants) | 14 | 14 | 14
  Transforming growth factor (TGF)-beta-1 | -0.199 (0.2853) | -0.465 (0.2884) | -0.077 (0.2521)
  CCL3: number analyzed (Participants) | 14 | 14 | 14
  CCL3 | -0.168 (0.4852) | -0.171 (0.5503) | 0.247 (0.7508)
  CX3CL1: number analyzed (Participants) | 14 | 14 | 14
  CX3CL1 | 0.346 (0.4784) | 0.458 (0.4269) | 0.012 (0.2771)
  CCL4: number analyzed (Participants) | 14 | 14 | 14
  CCL4 | -0.187 (0.3558) | -0.085 (0.5211) | 0.204 (0.4349)
  Membrane cofactor protein (MCP)-4: number analyzed (Participants) | 14 | 14 | 14
  Membrane cofactor protein (MCP)-4 | -0.627 (0.7270) | -0.860 (0.6659) | -0.116 (0.6018)
  MCP-3: number analyzed (Participants) | 14 | 14 | 14
  MCP-3 | -0.418 (0.8078) | -0.676 (0.5462) | -0.229 (0.7573)
  MCP-1: number analyzed (Participants) | 14 | 14 | 14
  MCP-1 | 0.053 (0.4337) | 0.108 (0.3722) | -0.081 (0.3836)
  MCP-2: number analyzed (Participants) | 14 | 14 | 14
  MCP-2 | -0.204 (0.2714) | -0.552 (0.3286) | -0.007 (0.2398)
  IL-1ra: number analyzed (Participants) | 14 | 14 | 14
  IL-1ra | -0.295 (0.4298) | -0.234 (0.6936) | -0.128 (0.6599)
  IL-6RA: number analyzed (Participants) | 14 | 14 | 14
  IL-6RA | -0.162 (0.2087) | -0.274 (0.1833) | -0.022 (0.1817)
  Tumor necrosis factor-related apoptosis-inducing ligand (TRAIL): number analyzed (Participants) | 14 | 14 | 14
  Tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) | -0.062 (0.2606) | -0.283 (0.2998) | 0.086 (0.2172)
  TNF-related weak inducer of apoptosis (TWEAK): number analyzed (Participants) | 14 | 14 | 14
  TNF-related weak inducer of apoptosis (TWEAK) | -0.057 (0.2239) | -0.157 (0.1705) | 0.099 (0.1471)
  EN-RAGE: number analyzed (Participants) | 14 | 14 | 14
  EN-RAGE | -0.175 (0.6414) | -0.383 (0.9149) | 0.175 (0.7755)
  P-selectin glycoprotein ligand-1 (PSGL-1): number analyzed (Participants) | 14 | 14 | 14
  P-selectin glycoprotein ligand-1 (PSGL-1) | -0.025 (0.2592) | -0.087 (0.1646) | -0.012 (0.1856)

5. Secondary Outcome: Percent-Change From Baseline in T-cell Lymphocyte Subset Populations at Week 12
Description: Mean percent changes from baseline at Week 12 in T-cell lymphocyte subset populations (CD3+ T cells, CD4+ T cells, CD8+ T cells, NK cells, B cells) are presented. Baseline is defined as the last observation on or prior to day of first dose (Day 1).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Percent change
  T-cells TBNK Screening (%): number analyzed (Participants) | 14 | 12 | 15
  T-cells TBNK Screening (%) | -0.2 (5.25) | 3.6 (6.65) | 1.7 (3.69)
  T-cells TBNK Screening (absolute): number analyzed (Participants) | 14 | 12 | 15
  T-cells TBNK Screening (absolute) | -14.5 (19.50) | 14.2 (43.43) | 1.5 (29.10)
  T lymphocytes CD3+CD4 (%): number analyzed (Participants) | 14 | 12 | 15
  T lymphocytes CD3+CD4 (%) | 1.4 (7.18) | 6.7 (11.73) | 5.6 (7.96)
  T lymphocytes CD3+CD4 (absolute): number analyzed (Participants) | 14 | 12 | 15
  T lymphocytes CD3+CD4 (absolute) | -13.2 (20.06) | 17.1 (41.66) | 5.2 (29.79)
  T lymphocytes CD3+CD8 (%): number analyzed (Participants) | 14 | 12 | 15
  T lymphocytes CD3+CD8 (%) | -0.7 (12.22) | 3.2 (10.59) | -1.6 (8.75)
  T lymphocytes CD3+CD8 (absolute): number analyzed (Participants) | 14 | 12 | 15
  T lymphocytes CD3+CD8 (absolute) | -15.1 (22.19) | 16.2 (54.75) | -1.1 (33.17)
  B-cells TBNK Screening (%): number analyzed (Participants) | 14 | 12 | 15
  B-cells TBNK Screening (%) | 35.5 (41.18) | 42.4 (37.49) | 7.8 (23.69)
  B-cells TBNK Screening (absolute): number analyzed (Participants) | 14 | 12 | 15
  B-cells TBNK Screening (absolute) | 18.3 (52.71) | 55.0 (59.81) | 7.7 (39.19)
  NK Cells TBNK Screening (%): number analyzed (Participants) | 14 | 12 | 15
  NK Cells TBNK Screening (%) | -27.3 (40.12) | -55.9 (24.04) | -15.2 (28.64)
  NK Cells TBNK Screening (absolute): number analyzed (Participants) | 14 | 12 | 15
  NK Cells TBNK Screening (absolute) | -40.0 (29.41) | -53.2 (26.96) | -17.9 (26.81)

6. Secondary Outcome: Response Based on at Least 4 Points Improvement in the Severity of Peak Pruritus Numerical Rating Scale (NRS) From Baseline and Changes From Baseline in Immunohistochemistry (IHC) and Gene Expression Biomarkers in Lesional Skin
Description: PP-NRS assesses the severity of itch (pruritus) due to AD. Participants were asked to assess their worst itching due to AD on an NRS anchored by the terms "no itch" (0) and "worst itch imaginable" (10). Participants who withdrew from the study were counted as non-responder. Spearman correlation coefficient was calculated to assess the relationship between PP-NRS CFB and fold CFB of IHC and gene expression biomarkers.
Time Frame: Baseline, Week 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and had response based on at least 4-points improvement from baseline in the severity of PP-NRS. Number Analyzed refers to the number of participants evaluable for each category.
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Spearman correlation coefficient
  CD11C | 0.242 | 0.484 | 0.439
  FC Epsilon R1 | 0.474 | 0.464 | 0.238
  CD3 | 0.438 | 0.408 | 0.151
  Macrophage mannose receptor 1 | 0.396 | 0.162 | -0.134
  S100A9 | 0.390 | 0.529 | 0.334
  S100A8 | 0.365 | 0.510 | 0.413
  KRT16 | 0.313 | 0.486 | 0.522
  S100A12 | 0.238 | 0.454 | 0.460
  CCL18 | 0.395 | 0.410 | 0.365

7. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of 'Clear' or 'Almost Clear' and >=2 Points Improvement From Baseline at Week 2, 4, 8 and 12
Description: The IGA of AD is scored on a 5-point scale (0-4), reflecting a global consideration of the erythema, induration and scaling. The overall severity of AD was assessed according to the 5-point scale: 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, and 4=Severe. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number Analyzed in each row refers to the number of participants measured and analyzed for each parameter at the specified visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Percentage of participants
  Week 2: number analyzed (Participants) | 16 | 13 | 16
  Week 2 | 0 [0.0 to 0.0] | 7.7 [0.0 to 22.2] | 0 [0.0 to 0.0]
  Week 4: number analyzed (Participants) | 15 | 14 | 15
  Week 4 | 26.7 [4.3 to 49.0] | 35.7 [10.6 to 60.8] | 0 [0.0 to 0.0]
  Week 8: number analyzed (Participants) | 15 | 14 | 15
  Week 8 | 26.7 [4.3 to 49.0] | 64.3 [39.2 to 89.4] | 0 [0.0 to 0.0]
  Week 12 | 25.0 [3.8 to 46.2] | 57.1 [31.2 to 83.1] | 0 [0.0 to 0.0]

8. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response ≥ 75% Improvement From Baseline Week 2, 4, 8 and 12
Description: The EASI quantifies the severity of AD based on both severity of lesion clinical signs and the percent of body surface area (BSA) affected. The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of AD. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline, Week 2, 4, 8, and 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Percentage of participants
  Week 2: number analyzed (Participants) | 16 | 13 | 16
  Week 2 | 6.3 [0.0 to 18.1] | 38.5 [12.0 to 64.9] | 0 [0.0 to 0.0]
  Week 4: number analyzed (Participants) | 15 | 14 | 15
  Week 4 | 46.7 [21.4 to 71.9] | 50.0 [23.8 to 76.2] | 0 [0.0 to 0.0]
  Week 8: number analyzed (Participants) | 15 | 14 | 15
  Week 8 | 46.7 [21.4 to 71.9] | 78.6 [57.1 to 100.0] | 0 [0.0 to 0.0]
  Week 12 | 43.8 [19.4 to 68.1] | 78.6 [57.1 to 100.0] | 0 [0.0 to 0.0]

9. Secondary Outcome: Percentage of Participants With >=4 Points at Baseline and Achieving >=4 Points Improvement From Baseline in Numeric Rating Scale for Severity of Pruritus (PP-NRS) at Weeks 2, 4, 8 and 12
Description: PP-NRS assesses the severity of itch (pruritus) due to AD. Participants were asked to assess their worst itching due to AD on an NRS anchored by the terms "no itch" (0) and "worst itch imaginable" (10). Higher scores indicated worse itch. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Percentage of participants
  Week 2 | 25.0 [3.8 to 46.2] | 57.1 [31.2 to 83.1] | 6.3 [0.0 to 18.1]
  Week 4: number analyzed (Participants) | 15 | 14 | 15
  Week 4 | 53.3 [28.1 to 78.6] | 64.3 [39.2 to 89.4] | 0 [0.0 to 0.0]
  Week 8: number analyzed (Participants) | 15 | 14 | 15
  Week 8 | 46.7 [21.4 to 71.9] | 64.3 [39.2 to 89.4] | 13.3 [0.0 to 30.5]
  Week 12: number analyzed (Participants) | 14 | 14 | 16
  Week 12 | 35.7 [10.6 to 60.8] | 64.3 [39.2 to 89.4] | 6.3 [0.0 to 18.1]

10. Secondary Outcome: Percentage of Participants Achieving EASI Response ≥ 90% Improvement From Baseline at Week 2, 4, 8 and 12
Description: The EASI quantifies the severity of AD based on both severity of lesion clinical signs and the percent of BSA affected. The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of AD. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline to Week 2, 4, 8 and 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Percentage of participants
  Week 2: number analyzed (Participants) | 16 | 13 | 16
  Week 2 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Week 4: number analyzed (Participants) | 15 | 14 | 15
  Week 4 | 20.0 [0.0 to 40.2] | 28.6 [4.9 to 52.2] | 0 [0.0 to 0.0]
  Week 8: number analyzed (Participants) | 15 | 14 | 15
  Week 8 | 20.0 [0.0 to 40.2] | 57.1 [31.2 to 83.1] | 0 [0.0 to 0.0]
  Week 12 | 37.5 [13.8 to 61.2] | 50.0 [23.8 to 76.2] | 0 [0.0 to 0.0]

11. Secondary Outcome: Percentage of Participants Achieving EASI Response ≥ 50% Improvement From Baseline at Week 2, 4, 8 and 12
Description: as for outcome 10
Time Frame: Baseline to Week 2, 4, 8 and 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number Analyzed in each row refers to the number of participants measured and analyzed for each parameter at specified visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Percentage of participants
  Week 2: number analyzed (Participants) | 16 | 13 | 16
  Week 2 | 37.5 [13.8 to 61.2] | 61.5 [35.1 to 88.0] | 12.5 [0.0 to 28.7]
  Week 4: number analyzed (Participants) | 15 | 14 | 15
  Week 4 | 66.7 [42.8 to 90.5] | 100.0 [100.0 to 100.0] | 6.7 [0.0 to 19.3]
  Week 8: number analyzed (Participants) | 15 | 14 | 15
  Week 8 | 53.3 [28.1 to 78.6] | 100.0 [100.0 to 100.0] | 6.7 [0.0 to 19.3]
  Week 12 | 68.8 [46.0 to 91.5] | 92.9 [79.4 to 100.0] | 18.8 [0.0 to 37.9]

12. Secondary Outcome: Percent Change From Baseline in Percentage Body Surface Area (BSA) at Week 2, 4, 8 and 12
Description: BSA efficacy is derived from the sum of the BSA in handprints across 4 body regions assessed as part of the EASI assessment. Handprint refers to that of each individual participant for their own measurement. The BSA efficacy ranges from 0 to 100%, with higher values representing greater severity of AD. The percentage BSA ranges from 0 to 100, with higher scores representing greater severity of AD. Since the scalp, palms, and soles were excluded from the BSA (efficacy) assessment, the maximum possible percentage BSA was less than 100.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Percent change
  Week 2: number analyzed (Participants) | 16 | 13 | 16
  Week 2 | -9.6 (12.06) | -17.3 (13.78) | 4.0 (17.25)
  Week 4: number analyzed (Participants) | 15 | 14 | 14
  Week 4 | -18.7 (15.70) | -23.8 (14.19) | 2.1 (18.35)
  Week 8: number analyzed (Participants) | 15 | 14 | 14
  Week 8 | -18.7 (20.96) | -28.3 (16.84) | 0.2 (21.59)
  Week 12: number analyzed (Participants) | 15 | 14 | 15
  Week 12 | -22.0 (19.03) | -28.3 (16.95) | -0.2 (23.20)

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. TEAEs were AEs that occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator.
Time Frame: Baseline to 16 weeks
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Participants
  All-causality TEAEs | 10 | 7 | 8
  Treatment-related TEAEs | 6 | 5 | 3

14. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Treatment-related SAEs were determined by the investigator.
Time Frame: Baseline to 16 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Participants
  All-causality SAEs | 0 | 0 | 1
  Treatment-related SAEs | 0 | 0 | 1

15. Secondary Outcome: Number of Participants Who Discontinued From the Study Due to TEAEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. TEAEs were AEs that occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator.
Time Frame: Baseline to 16 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Participants
  All-causality TEAEs | 2 | 1 | 2
  Treatment-related TEAEs | 2 | 1 | 1

16. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory tests included hematology (including coagulation panel), clinical chemistry, lipid profile panel, and routine urinalysis. LLN is lower limit of normal. ULN is upper limit of normal.
Time Frame: Baseline to 16 weeks
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number of Participants Analyzed refers to the number of participants who were evaluable for this outcome measure. Number analyzed refers to the number of participants with at least one observation of the given laboratory test.
Measure: Number; unit: Participants
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Participants
  Hemoglobin (g/dL) <0.8*LLN | 1 | 0 | 0
  Hematocrit (%) < 0.8*LLN | 1 | 0 | 0
  Erythrocytes (10^6/mm3) < 0.8*LLN | 1 | 0 | 0
  Reticulocytes (10^3/mm3) < 0.5*LLN | 1 | 0 | 0
  Platelets (10^3/mm3) < 0.5*LLN | 1 | 0 | 0
  Reticulocytes/Erythrocytes (%) > 1.5*ULN | 1 | 0 | 0
  Leukocytes (10^3/mm3) < 0.6*LLN | 1 | 0 | 0
  Lymphocytes (10^3/mm3) < 0.8*LLN | 2 | 0 | 0
  Lymphocytes/Leukocytes (%) < 0.8*LLN | 3 | 0 | 1
  Lymphocytes/Leukocytes (%) > 1.2*ULN | 0 | 1 | 0
  Neutrophils (10^3/mm3) < 0.8*LLN | 1 | 3 | 0
  Neutrophils/Leukocytes (%) < 0.8*LLN | 0 | 2 | 2
  Basophils/Leukocytes (%) > 1.2*ULN | 1 | 1 | 2
  Eosinophils (10^3/mm3) > 1.2*ULN | 5 | 2 | 10
  Eosinophils/Leukocytes (%) > 1.2*ULN | 6 | 2 | 10
  Monocytes (10^3/mm3) > 1.2x ULN | 0 | 1 | 0
  Monocytes/Leukocytes (%) > 1.2*ULN | 1 | 3 | 0
  Prothrombin Time (sec) > 1.1*ULN | 1 | 0 | 0
  Bilirubin (mg/dL) > 1.5*ULN: number analyzed (Participants) | 16 | 14 | 15
  Bilirubin (mg/dL) > 1.5*ULN | 0 | 1 | 0
  Indirect Bilirubin (mg/dL) > 1.5*ULN: number analyzed (Participants) | 16 | 14 | 15
  Indirect Bilirubin (mg/dL) > 1.5*ULN | 0 | 1 | 0
  Aspartate Aminotransferase (U/L) > 3.0*ULN: number analyzed (Participants) | 16 | 14 | 15
  Aspartate Aminotransferase (U/L) > 3.0*ULN | 0 | 1 | 0
  Alanine Aminotransferase (U/L) > 3.0*ULN: number analyzed (Participants) | 16 | 14 | 15
  Alanine Aminotransferase (U/L) > 3.0*ULN | 0 | 0 | 1
  Gamma Glutamyl Transferase (U/L) > 3.0*ULN: number analyzed (Participants) | 16 | 14 | 15
  Gamma Glutamyl Transferase (U/L) > 3.0*ULN | 1 | 0 | 0
  Lactate Dehydrogenase (U/L) > 3.0*ULN: number analyzed (Participants) | 16 | 14 | 15
  Lactate Dehydrogenase (U/L) > 3.0*ULN | 0 | 1 | 0
  Creatinine (mg/dL) > 1.3*ULN: number analyzed (Participants) | 16 | 14 | 15
  Creatinine (mg/dL) > 1.3*ULN | 1 | 0 | 0
  Urate (mg/dL) > 1.2*ULN: number analyzed (Participants) | 16 | 14 | 15
  Urate (mg/dL) > 1.2*ULN | 1 | 1 | 0
  Potassium (mEq/L) < 0.9*LLN: number analyzed (Participants) | 16 | 14 | 15
  Potassium (mEq/L) < 0.9*LLN | 1 | 1 | 0
  Bicarbonate (mEq/L) > 1.1*ULN: number analyzed (Participants) | 16 | 14 | 15
  Bicarbonate (mEq/L) > 1.1*ULN | 0 | 1 | 0
  Creatine Kinase (U/L) > 2.0*ULN: number analyzed (Participants) | 16 | 14 | 15
  Creatine Kinase (U/L) > 2.0*ULN | 1 | 3 | 2
  Cholesterol (mg/dL) > 1.3*ULN: number analyzed (Participants) | 16 | 14 | 15
  Cholesterol (mg/dL) > 1.3*ULN | 0 | 0 | 1
  Ketones ≥ 1: number analyzed (Participants) | 16 | 14 | 15
  Ketones ≥ 1 | 0 | 2 | 0
  URINE Protein ≥ 1: number analyzed (Participants) | 16 | 14 | 15
  URINE Protein ≥ 1 | 0 | 1 | 1
  URINE Hemoglobin ≥ 1: number analyzed (Participants) | 16 | 14 | 15
  URINE Hemoglobin ≥ 1 | 2 | 2 | 0
  Leukocyte Esterase ≥ 1: number analyzed (Participants) | 16 | 14 | 15
  Leukocyte Esterase ≥ 1 | 5 | 3 | 1
  URINE Leukocytes (Scalar) ≥ 20: number analyzed (Participants) | 15 | 11 | 14
  URINE Leukocytes (Scalar) ≥ 20 | 2 | 0 | 0
  Hyaline Casts (/LPF) > 1: number analyzed (Participants) | 2 | 3 | 0
  Hyaline Casts (/LPF) > 1 | 2 | 1 |

17. Other Pre Specified Outcome: Change From Baseline in Erythrocytes at Week 2, 4, 8 and 12
Description: Clinical laboratory tests including red blood cell (erythrocytes) were performed at Week 2, 4, 8, and 12 by collecting blood samples and performing the corresponding analysis per the laboratory manual. Fasting was only required prior to labs that included the lipid profile panel.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^6 cells/mm^3
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
10^6 cells/mm^3
  Week 2: number analyzed (Participants) | 14 | 14 | 15
  Week 2 | -0.12 (0.212) | -0.21 (0.305) | -0.10 (0.242)
  Week 4: number analyzed (Participants) | 14 | 14 | 14
  Week 4 | -0.16 (0.279) | -0.19 (0.266) | -0.11 (0.274)
  Week 8: number analyzed (Participants) | 13 | 13 | 14
  Week 8 | -0.21 (0.301) | -0.35 (0.424) | -0.02 (0.246)
  Week 12: number analyzed (Participants) | 15 | 14 | 15
  Week 12 | -0.35 (0.376) | -0.47 (0.434) | 0.07 (0.183)

18. Other Pre Specified Outcome: Change From Baseline in Reticulocytes at Week 2, 4, 8 and 12
Description: Clinical laboratory tests including reticulocytes were performed at Week 2, 4, 8, and 12 by collecting blood samples and performing the corresponding analysis per the laboratory manual. Fasting was only required prior to labs that included the lipid profile panel.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^3 cells/mm^3
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
10^3 cells/mm^3
  Week 2: number analyzed (Participants) | 14 | 14 | 15
  Week 2 | -15.43 (23.177) | -25.14 (28.057) | 5.33 (12.199)
  Week 4: number analyzed (Participants) | 14 | 14 | 14
  Week 4 | -11.64 (27.845) | -20.86 (28.710) | 1.86 (16.209)
  Week 8: number analyzed (Participants) | 13 | 13 | 14
  Week 8 | -9.31 (15.997) | -13.23 (18.682) | 0.07 (15.345)
  Week 12: number analyzed (Participants) | 15 | 14 | 15
  Week 12 | -5.07 (16.615) | -7.64 (28.169) | 4.33 (20.318)

19. Other Pre Specified Outcome: Change From Baseline in Platelet Counts at Week 2, 4, 8 and 12
Description: Clinical laboratory tests including platelet counts were performed at Week 2, 4, 8, and 12 by collecting blood samples and performing the corresponding analysis per the laboratory manual. Fasting was only required prior to labs that included the lipid profile panel.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^3 cells/mm^3
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
10^3 cells/mm^3
  Week 2: number analyzed (Participants) | 14 | 13 | 15
  Week 2 | -72.86 (93.413) | -53.23 (28.176) | 12.87 (51.582)
  Week 4: number analyzed (Participants) | 14 | 14 | 14
  Week 4 | -89.79 (123.180) | -93.29 (36.123) | 11.79 (33.025)
  Week 8: number analyzed (Participants) | 13 | 13 | 14
  Week 8 | -68.15 (102.846) | -71.38 (44.925) | 5.79 (28.917)
  Week 12: number analyzed (Participants) | 15 | 14 | 15
  Week 12 | -59.00 (104.408) | -65.79 (42.600) | 5.47 (34.620)

20. Other Pre Specified Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP) at Week 2, 4, 8 and 12
Description: Clinical laboratory tests including hs-CRP were performed at Week 2, 4, 8, and 12 by collecting blood samples and performing the corresponding analysis per the laboratory manual. Fasting was only required prior to labs that included the lipid profile panel.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
milligrams per deciliter
  Week 2: number analyzed (Participants) | 15 | 14 | 15
  Week 2 | -0.26 (0.431) | -0.07 (0.147) | -0.13 (1.538)
  Week 4: number analyzed (Participants) | 15 | 14 | 14
  Week 4 | -0.24 (0.376) | -0.09 (0.217) | -0.43 (1.283)
  Week 8: number analyzed (Participants) | 14 | 14 | 14
  Week 8 | -0.19 (0.287) | 0.03 (0.253) | -0.42 (1.182)
  Week 12: number analyzed (Participants) | 16 | 14 | 15
  Week 12 | -0.15 (0.368) | 0.01 (0.254) | -0.40 (1.114)

21. Other Pre Specified Outcome: Change From Baseline in Interleukin 6 at Week 2, 4, 8 and 12
Description: Clinical laboratory tests including interleukin were performed at Week 2, 4, 8, and 12 by collecting blood samples and performing the corresponding analysis per the laboratory manual. Fasting was only required prior to labs that included the lipid profile panel.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
picograms per milliliter
  Week 2: number analyzed (Participants) | 15 | 13 | 14
  Week 2 | -0.02 (2.732) | -0.11 (7.021) | -0.44 (2.797)
  Week 4: number analyzed (Participants) | 15 | 14 | 14
  Week 4 | 0.16 (2.533) | -0.85 (5.045) | -1.83 (6.034)
  Week 8: number analyzed (Participants) | 13 | 13 | 14
  Week 8 | 0.19 (1.391) | 0.15 (5.728) | -3.52 (8.228)
  Week 12: number analyzed (Participants) | 16 | 14 | 15
  Week 12 | -0.23 (2.712) | -0.19 (5.305) | -2.59 (6.339)

22. Other Pre Specified Outcome: Change From Baseline in Erythropoietin at Week 2, 4, 8 and 12
Description: Clinical laboratory tests including erythropoietin were performed at Week 2, 4, 8, and 12 by collecting blood samples and performing the corresponding analysis per the laboratory manual. Fasting was only required prior to labs that included the lipid profile panel.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milliunits per milliliter
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
milliunits per milliliter
  Week 2: number analyzed (Participants) | 15 | 14 | 14
  Week 2 | 5.38 (7.042) | 15.78 (29.596) | 0.59 (7.412)
  Week 4: number analyzed (Participants) | 15 | 14 | 14
  Week 4 | 5.30 (6.286) | 14.60 (30.438) | 0.35 (8.294)
  Week 8: number analyzed (Participants) | 14 | 13 | 14
  Week 8 | 7.84 (8.305) | 34.12 (58.113) | -1.99 (8.101)
  Week 12: number analyzed (Participants) | 16 | 14 | 15
  Week 12 | 7.86 (15.831) | 54.08 (136.613) | -3.11 (6.391)

23. Other Pre Specified Outcome: Change From Baseline in Thrombopoietin at Week 2, 4, 8 and 12
Description: Clinical laboratory tests including thrombopoietin were performed at Week 2, 4, 8, and 12 by collecting blood samples and performing the corresponding analysis per the laboratory manual. Fasting was only required prior to labs that included the lipid profile panel.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Picograms per milliliter (pg/mL)
  Week 2: number analyzed (Participants) | 15 | 14 | 14
  Week 2 | 38.33 (61.921) | 47.64 (38.472) | 13.29 (31.665)
  Week 4: number analyzed (Participants) | 15 | 14 | 14
  Week 4 | 107.93 (274.324) | 103.07 (136.964) | -9.36 (31.030)
  Week 8: number analyzed (Participants) | 14 | 13 | 14
  Week 8 | 26.93 (49.260) | 76.54 (116.433) | 4.57 (33.073)
  Week 12: number analyzed (Participants) | 15 | 14 | 15
  Week 12 | 30.93 (53.723) | 89.57 (201.700) | -7.00 (30.166)

24. Other Pre Specified Outcome: Change From Baseline in Night Time Itch Scale Score at Week 2, 4, 8 and 12
Description: The severity and frequency of itch (pruritus) during the night due to AD was assessed using the Night Time Itch Scale Score. Participants assessed their worst itching due to AD during their most recent night's sleep on an NRS anchored by the terms "no itch" (0) and "worst itch imaginable" (10). Higher scores indicated worse itch. The frequency of itch was assessed using a 5-point qualitative scale, with responses including "Never", "Rarely", "Sometimes", "Often" and "Almost Always".
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
Number analyzed (Participants) | 16 | 14 | 16
Units on a scale
  NRS01-Severity of Night Time Itch Week 2: number analyzed (Participants) | 16 | 14 | 15
  NRS01-Severity of Night Time Itch Week 2 | -2.4 (2.16) | -4.6 (2.79) | -0.3 (1.83)
  NRS01-Severity of Night Time Itch Week 4: number analyzed (Participants) | 15 | 14 | 13
  NRS01-Severity of Night Time Itch Week 4 | -4.4 (3.38) | -4.9 (3.52) | -1.1 (2.53)
  NRS01-Severity of Night Time Itch Week 8: number analyzed (Participants) | 15 | 14 | 13
  NRS01-Severity of Night Time Itch Week 8 | -3.5 (4.14) | -5.5 (3.52) | -0.8 (2.85)
  NRS01-Severity of Night Time Itch Week 12: number analyzed (Participants) | 13 | 14 | 14
  NRS01-Severity of Night Time Itch Week 12 | -3.4 (3.80) | -4.8 (3.77) | -1.1 (2.46)
  NRS01-Frequency of Night Time Itch Week 2: number analyzed (Participants) | 16 | 14 | 15
  NRS01-Frequency of Night Time Itch Week 2 | -0.8 (0.91) | -2.1 (1.14) | -0.2 (1.08)
  NRS01-Frequency of Night Time Itch Week 4: number analyzed (Participants) | 15 | 14 | 13
  NRS01-Frequency of Night Time Itch Week 4 | -1.8 (1.08) | -2.5 (1.09) | -0.6 (1.12)
  NRS01-Frequency of Night Time Itch Week 8: number analyzed (Participants) | 15 | 14 | 13
  NRS01-Frequency of Night Time Itch Week 8 | -1.4 (1.35) | -2.7 (1.14) | -0.6 (1.39)
  NRS01-Frequency of Night Time Itch Week 12: number analyzed (Participants) | 13 | 14 | 14
  NRS01-Frequency of Night Time Itch Week 12 | -1.2 (1.21) | -2.5 (1.45) | -0.4 (1.22)

25. Other Pre Specified Outcome: Plasma PF-04965842 Concentration
Description: Pharmacokinetic (PK) samples were collected at Week 4 and 12 for measurement of plasma concentration of PF-04965842.
Time Frame: Day 29 Hour 0 (prior to dosing) and 30 miniute post-dose, Day 85 30 minute and Hour 4 post-dose
Population: The PK analysis included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number Analyzed in each row refers to the number of participants with the corresponding PK parameter measured and analyzed at specified visit.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD
Number analyzed (Participants) | 16 | 14
nanogram per milliliter (ng/mL)
  Day 29 Hour 0: number analyzed (Participants) | 11 | 13
  Day 29 Hour 0 | 14.77 (29.293) | 135.7 (272.53)
  Day 29 30 minute: number analyzed (Participants) | 14 | 12
  Day 29 30 minute | 266.6 (381.11) | 802.7 (1128.2)
  Day 85 30 minute: number analyzed (Participants) | 14 | 13
  Day 85 30 minute | 617.6 (588.85) | 792.2 (1013.9)
  Day 85 Hour 4: number analyzed (Participants) | 14 | 12
  Day 85 Hour 4 | 433.0 (255.44) | 1147 (580.56)

26. Other Pre Specified Outcome: Plasma PF-06471658 (M1) Concentration
Description: PK samples were collected at Week 4 and 12 for measurement of plasma concentration of abrocitinib's metabolite PF-06471658 (M1).
Time Frame: Day 29 Hour 0 (prior to dosing) and 30 miniute post-dose, Day 85 30 minute and Hour 4 post-dose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD
Number analyzed (Participants) | 16 | 14
ng/mL
  Day 29 Hour 0: number analyzed (Participants) | 10 | 13
  Day 29 Hour 0 | 2.588 (3.4071) | 23.13 (47.649)
  Day 29 30 minute: number analyzed (Participants) | 12 | 13
  Day 29 30 minute | 65.82 (137.66) | 95.54 (108.21)
  Day 85 30 minute: number analyzed (Participants) | 14 | 13
  Day 85 30 minute | 92.51 (80.717) | 65.03 (51.765)
  Day 85 Hour 4: number analyzed (Participants) | 14 | 12
  Day 85 Hour 4 | 82.84 (70.532) | 104.9 (80.782)

27. Other Pre Specified Outcome: Plasma PF-07055087 (M2) Concentration
Description: PK samples were collected at Week 4 and 12 for measurement of plasma concentration of abrocitinib's metabolite PF-07055087 (M2).
Time Frame: Day 29 Hour 0 (prior to dosing) and 30 miniute post-dose, Day 85 30 minute and Hour 4 post-dose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD
Number analyzed (Participants) | 16 | 14
ng/mL
  Day 29 Hour 0: number analyzed (Participants) | 7 | 9
  Day 29 Hour 0 | 9.933 (22.629) | 23.86 (40.798)
  Day 29 30 minute: number analyzed (Participants) | 10 | 11
  Day 29 30 minute | 42.89 (66.789) | 73.84 (75.245)
  Day 85 30 minute: number analyzed (Participants) | 13 | 13
  Day 85 30 minute | 77.56 (63.483) | 70.58 (67.136)
  Day 85 Hour 4: number analyzed (Participants) | 14 | 12
  Day 85 Hour 4 | 100.0 (46.321) | 132.9 (69.048)

28. Other Pre Specified Outcome: Plasma PF-07054874 (M4) Concentration
Description: PK samples were collected at Week 4 and 12 for measurement of plasma concentration of abrocitinib's metabolites PF-07054874 (M4).
Time Frame: Day 29 Hour 0 (prior to dosing) and 30 miniute post-dose, Day 85 30 minute and Hour 4 post-dose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD
Number analyzed (Participants) | 16 | 14
ng/mL
  Day 29 Hour 0: number analyzed (Participants) | 14 | 13
  Day 29 Hour 0 | 16.10 (33.537) | 48.43 (83.563)
  Day 29 30 minute: number analyzed (Participants) | 15 | 13
  Day 29 30 minute | 63.76 (80.663) | 153.4 (163.23)
  Day 85 30 minute: number analyzed (Participants) | 14 | 13
  Day 85 30 minute | 149.9 (126.33) | 158.2 (174.55)
  Day 85 Hour 4: number analyzed (Participants) | 14 | 11
  Day 85 Hour 4 | 170.4 (68.419) | 268.2 (173.11)

ADVERSE EVENTS:
Time Frame: Baseline up to 16 weeks
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Abrocitinib 100 mg QD | Abrocitinib 200 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 1/16
Other Adverse Events (participants affected / at risk) | 10/16 | 7/14 | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abrocitinib 100 mg QD (N=16) | Abrocitinib 200 mg QD (N=14) | Placebo (N=16)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abrocitinib 100 mg QD (N=16) | Abrocitinib 200 mg QD (N=14) | Placebo (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood erythropoietin increased (Investigations) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Large intestinal polypectomy (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03915496/Prot_004.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT03915496/SAP_005.pdf